CLINICAL TRIAL: NCT04072939
Title: Study of the Incidence of Retinal Detachment After Lens Surgery in the Nearsighted
Brief Title: Retinal Detachment After Lens Surgery in the Nearsighted
Acronym: A09F0401
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2004/03
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Retinal Detachment; Lens Diseases; Short-Sighted
Keywords: Phacoemulsification
MeSH Terms: conditions — Retinal Detachment; Lens Diseases; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Single arm: dilated fundus exam
  Interventions: Other: Patients having had a lens surgery

INTERVENTIONS:
Other: Patients having had a lens surgery — Dilated fundus exam

SUMMARY:
This study aims to study the incidence of retinal detachment in the nearsighted myopic after phakoemulsification lens surgery and use of posterior chamber foldable soft implants with a follow-up of 5 years and preliminary results at 3 years.

DETAILED DESCRIPTION:
Major advances have been made in the field of lens surgery over the last 20 years which has significantly reduced the per and postoperative complications of this surgery. Retinal detachment remains the most feared complication of this surgery in the nearsighted.

There is currently an increasing popularity in the international ophthalmic community for the correction of ametropia, particularly nearsightedness, by ablation of the non-cataracted lens, referred to as refractive lensectomy. However, no recent study reports the complications of this procedure with the use of modern surgical techniques.

This study aims to study the incidence of retinal detachment in the nearsighted myopic after phakoemulsification lens surgery and use of posterior chamber foldable soft implants with a follow-up of 5 years and preliminary results at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Male or female aged 20 to 60 included.
* Myopia: axile, united or bilateral.
* Degree of myopia: Axial length of the eye to be operated ≥ 26 mm, measured by ultrasound A or B.
* Preoperative visual acuity of the eye to be operated ≥ 0.2.
* Crystalline eye to operate natural: clear or opacified (allowed: cataract complicating a myopic implant and cataract after corneal refractive surgery.

Exclusion Criteria:

* History of retinal detachment on the eye to be operated or the eye to help.
* History of glaucoma of the eye to operate.
* intraocular pressure of the eye to operate ≥ 21 mmHg.
* History of diabetic retinopathy.
* History of anterior or posterior intraocular inflammation in the year preceding surgery.
* History of vitreoretinal syndrome (Stickler's disease ...).
* Unstable systemic pathology in the month preceding the preoperative check-up (Visit 1) (example: uncontrolled hypertension, diabetes with abnormal glycemia, thyroid disorders, uncontrolled autoimmune diseases, etc.) or deemed by the investigator to be incompatible with the study (example: hepatic or renal insufficiency, all severe chronic organic diseases: metabolic, endocrine, neoplastic, hematological, etc., severe psychiatric diseases).
* Pregnancy, breastfeeding.
* History of filter surgery of the eye to be operated.
* History of vitreoretinal surgery of the eye to be operated (authorized after Day 0).
* Patient unable to understand the instructions of the study or not likely to comply with the course of the study and treatment.
* Participation in another clinical trial in the month preceding the start of this study, at the same time as this study.
* Patient not covered by the French social security system.
* Major patient under guardianship.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Strong myopic patients with lens surgery
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2005-05-31 (Actual); Primary Completion 2006-08-31 (Actual); Study Completion 2006-08-31 (Actual)

PRIMARY OUTCOMES:
Posterior detachment of vitreous yes/no | Preoperative time
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Posterior detachment of vitreous yes/no | 1 day after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Posterior detachment of vitreous yes/no | 1 week after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Posterior detachment of vitreous yes/no | 1 month after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Posterior detachment of vitreous yes/no | 3 months after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
lesions of the retinal periphery yes/no | Preoperative time
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
lesions of the retinal periphery yes/no | 1 day after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
lesions of the retinal periphery yes/no | 1 week after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
lesions of the retinal periphery yes/no | 1 month after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
lesions of the retinal periphery yes/no | 3 months after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Argon laser treatment scars yes/no | Preoperative time
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Argon laser treatment scars yes/no | 1 day after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Argon laser treatment scars yes/no | 1 week after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Argon laser treatment scars yes/no | 1 month after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Argon laser treatment scars yes/no | 3 months after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
tabby appearance without atrophy yes/no | Preoperative time
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
tabby appearance without atrophy yes/no | 1 day after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
tabby appearance without atrophy yes/no | 1 week after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
tabby appearance without atrophy yes/no | 1 month after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
tabby appearance without atrophy yes/no | 3 months after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Presence of eye anomaly yes/no (myopic conus, Bruch's membrane breaks, deep chorioretinal atrophic cupboard with punch, deep choroidal atrophic cupboard showing sclera to bare) | Preoperative time
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Presence of eye anomaly yes/no (myopic conus, Bruch's membrane breaks, deep chorioretinal atrophic cupboard with punch, deep choroidal atrophic cupboard showing sclera to bare) | 1 day after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Presence of eye anomaly yes/no (myopic conus, Bruch's membrane breaks, deep chorioretinal atrophic cupboard with punch, deep choroidal atrophic cupboard showing sclera to bare) | 1 week after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Presence of eye anomaly yes/no (myopic conus, Bruch's membrane breaks, deep chorioretinal atrophic cupboard with punch, deep choroidal atrophic cupboard showing sclera to bare) | 1 month after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.
Presence of eye anomaly yes/no (myopic conus, Bruch's membrane breaks, deep chorioretinal atrophic cupboard with punch, deep choroidal atrophic cupboard showing sclera to bare) | 3 months after surgery
  With dilated fundus exam: the pupil will be dilated by instillation of a mydriatic eye drop. The bottom of the eye and the peripheral retina will be examined with a slit lamp with a Superfield lens or a glass with 3 mirrors.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph COLIN, Pr, Principal Investigator — Bordeaux University hsopital

IPD SHARING:
Plan to Share IPD: No